CLINICAL TRIAL: NCT00754143
Title: A Randomized, Double-blind, Placebo-Controlled, Phase 1 Study of Safety, Pharmacokinetics and Pharmacodynamics of FG-3019 in Subjects With Type 1 or Type 2 Diabetes Mellitus and Diabetic Nephropathy on Background ACEi and/or ARB Therapy
Brief Title: Phase 1 Study of FG-3019 in Subjects With Type 1 or Type 2 Diabetes Mellitus and Diabetic Nephropathy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyntra Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FGCL-3019-029
Record Dates: First submitted 2008-09-15; First posted 2008-09-17 (Estimated); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Diabetes Mellitus; Diabetic Nephropathy
Keywords: Type 1 or Type 2 diabetes; proteinuria
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Nephropathies; Diabetes Mellitus, Type 2; Proteinuria | interventions — pamrevlumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Placebo Comparator): Placebo
  Interventions: Drug: FG-3019
- B (Experimental): FG-3019 5 mg/kg
  Interventions: Drug: FG-3019
- C (Experimental): FG-3019 10 mg/kg
  Interventions: Drug: FG-3019

INTERVENTIONS:
Drug: FG-3019 — Placebo every 2 weeks IV for all infusions
  Arms: A
Drug: FG-3019 — FG-3019 5 mg/kg every 2 weeks IV for all infusions
  Arms: B
Drug: FG-3019 — FG-3019 10 mg/kg IV for infusions on Days 1, 15, 29 and 57 and Placebo IV on Days 43 and 71
  Arms: C

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of two dosing regimens of FG-3019 administered over 12 weeks in patients with diabetic nephropathy and proteinuria on background angiotensin converting enzyme inhibitor (ACEi) and/or angiotensin II receptor antagonist (ARB) therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years, inclusive
2. Diagnosis of type 1 or type 2 diabetes according to American Diabetes Association (ADA) criteria
3. First morning urinary ACR >0.200 g/g
4. Receiving stable doses of ACEi and/or ARB therapy prior to Screening
5. Estimated glomerular filtration rate of ≥20 and <90 mL/min/1.73 m2
6. Willingness to maintain ACEi and/or ARB therapy, and any additional anti-hypertensive therapies to control blood pressure, at a stable dose
7. Maintenance of all additional antihypertensive medications, insulin, oral hypoglycemic agents, and cholesterol-lowering medications prior to randomization

Exclusion Criteria:

1. Female subjects who are pregnant or breastfeeding
2. Organ transplant recipient, previous dialysis, or non-diabetic renal disease other than benign cysts or anatomical variants
3. Any history of New York Heart Association (NYHA) class III/IV heart failure (HF)
4. Screening electrocardiogram showing acute, clinically significant findings including but not limited to ST depression
5. Recent history of serious heart problems (e.g. coronary artery bypass graft, cerebrovascular accident, or myocardial infarction)
6. History of cancer in the past 5 years, possibly excluding non-melanomatous skin cancer, localized bladder cancer, or in situ cervical cancer.
7. History of allergic or anaphylactic reaction to human, humanized, chimeric or murine monoclonal antibodies
8. Participation in other studies of investigational drugs at the time of Screening AND receipt of an investigational drug within 42 days prior to Screening
9. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2.5 times the upper limit of normal
10. Hemoglobin <10 g/dL
11. Positive for HIV (IgG) antibody

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2008-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of FG-3019 | 34 weeks

SECONDARY OUTCOMES:
Pharmacokinetic parameters | 34 weeks
Change from baseline in first morning urinary albumin creatinine ratio (ACR) | 6 weeks (10 mg/kg) or 10 weeks (5 mg/kg)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Birmingham, Alabama
  - Tempe, Arizona
  - La Mesa, California
  - Torrance, California
  - Kissimmee, Florida
  - Atlanta, Georgia
  - Springfield, Massachusetts
  - Omaha, Nebraska
  - Flushing, New York
  - New York, New York
  - Chapel Hill, North Carolina
  - Cleveland, Ohio
  - Portland, Oregon
  - Hershey, Pennsylvania
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Fairfax, Virginia